CLINICAL TRIAL: NCT05664074
Title: Post ERCP Pancreatitis Prophylaxis, Effectiveness of Rectal Indomethacin vs Intravenous Ketorolac in the Pediatric Population
Brief Title: Rectal Indomethacin vs Intravenous Ketorolac
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: David Vitale MD (Other)
Responsible Party: Sponsor-Investigator, David Vitale MD, Assistant Professor, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-0640
Record Dates: First submitted 2022-11-23; First posted 2022-12-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Post-ERCP Acute Pancreatitis
MeSH Terms: interventions — Ketorolac

STUDY DESIGN:
Intervention Model Description: This will be a prospective study where patients will be randomized into either rectal indomethacin or IV ketorolac.
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectal indomethacin (Experimental): Dosage based on subject's weight:
  >=50 kg, 100 mg; 30-49 kg, 50 mg; 10-29 kg, 25 mg
  Interventions: Drug: Rectal indomethacin
- IV ketorolac (Experimental): Dosage based on subject's weight: 0.5 mg/kg (maximum: 15 mg)
  Interventions: Drug: IV ketorolac

INTERVENTIONS:
Drug: Rectal indomethacin — Dosage based on subject's weight:
  >=50 kg, 100 mg; 30-49 kg, 50 mg; 10-29 kg, 25 mg
  Arms: Rectal indomethacin
Drug: IV ketorolac — Dosage based on subject's weight: 0.5 mg/kg (maximum: 15 mg)
  Arms: IV ketorolac

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) is an essential procedure that can be complicated by post-ERCP pancreatitis (PEP). Indomethacin and ketorolac are two medications used to prevent PEP. The main reason for this research study is to compare the effectiveness these drugs at reducing rates of PEP. There have been no studies comparing the effectiveness of these medications in preventing PEP in pediatric patients. You are being asked to take part in this research study because you are scheduled to have an ERCP as part of your medical care.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing ERCP (diagnostic or therapeutic with cannulation of the major or minor papilla)
* Age 6 month- 21 years old
* Does not meet exclusion criteria

Exclusion Criteria:

* < 10 kg
* Low risk subgroup: Biliary indication with history of prior biliary sphincterotomy.
* High risk for bleeding (Example: Planned liver biopsy)
* Gastrointestinal bleeding in previous 3 days
* Acute pancreatitis (within 3 days) at the time of ERCP
* Use of NSAIDs in the previous 5 days
* Peptic ulcer disease
* Acute kidney Injury or Known Chronic Kidney Disease per KDIGO
* Pregnancy (Pregnancy tests are administered prior to ERCP as standard of care)
* Lithium therapy
* Allergy to ketorolac or indomethacin
* Organ Dysfunction or SIRS

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 192 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Post-ERCP Pancreatitis | 2 weeks
  Number of patient who develop Post-ERCP Pancreatitis-
  Post ERCP Pancreatitis: A patient must have at least 2 of the following to establish a diagnosis of post ERCP pancreatitis:
  1. Characteristic physical exam findings- pain worse than admission per pain scales (please see point 2) and/or nausea
  2. Amylase (unit/L) or lipase(unit/L) greater than 3 times the age appropriate upper limit of normal.
     * Normal range of amylase (15-127 unit/L)
     * Normal range of lipase (12-50 unit/L)
  3. Confirmatory imaging (Ultrasound, CT or MRI) that suggests or demonstrates pancreatic inflammation

SECONDARY OUTCOMES:
Pain assessed by FLACC or NRS scoring post ERCP | 2 weeks
  A minimum of 3 pain assessments are to be completed by nursing staff/anesthesia during admission:
  Anesthesia/ PACU- initial pain assessment Evening-2100- pain assessment by RN Morning -0800- pain assessment by RN
  Face, Legs, Activity, Cry, and Consolability (FLACC) Pain scale for patients 0-5 years of age and patients unable to verbalize pain
  Numeric Rating Scale (NRS) Pain scale for patients 6 years old and above
  1. Mild- 0 to 3
  2. Moderate- 4 to 6
  3. Severe- 7 to 10
Laboratory markers associated PEP (Amylase and Lipase) | 2 weeks
  Amylase (unit/L) Lipase (unit/L)
Length of stay | 2 weeks
Severity of pancreatitis (mild, moderately severe, severe) | 2 weeks
  Severity of Acute Pancreatitis (AP): Severity of AP will be classified as mild, moderately severe, or severe in accordance with the NASPGHAN Classification system.
  1. Mild: "AP that is not associated with any organ failure, local or systemic complications, and usually resolves within the first week after presentation."
  2. Moderately Severe: "AP with either the development of transient organ failure/dysfunction (lasting no >48 hours) or development of local or systemic complications. Local complications would include development of (peri) or pancreatic complications including fluid collections or necrosis. Systemic complications would include exacerbation of previously diagnosed co-morbid disease (such as lung disease or kidney disease)."
  3. Severe: "AP with development of organ dysfunction per International pediatric sepsis consensus conference that persists >48 hours. Persistent organ failure may be single or multiple, and may develop beyond the first 48 hours of presentation."
C-Reactive Protein (CRP) level | 2 weeks
  Measured in mg/dL
Post-ERCP bleeding | 2 weeks
White Blood Cell | 2 weeks
  per/mcL
Red Blood Cell | 2 weeks
  per/mcL
Hemoglobin | 2 weeks
  gm/dL
Hematocrit | 2 weeks
MCV | 2 weeks
  fL
MCH | 2 weeks
  pg
MCHC | 2 weeks
  gm/dL
RDW | 2 weeks
PLATELET | 2 weeks
  per/mcL

CONTACTS AND LOCATIONS:
Overall Officials: David Vitale, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT05664074/SAP_000.pdf
  • Informed Consent Form (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT05664074/ICF_001.pdf